CLINICAL TRIAL: NCT02038088
Title: The Effect of General Anesthesia Immunosuppressive on Hepatitis B Virus Replication
Acronym: HBV
Status: Completed | Type: Observational
Sponsor: Lu KZ (Other)
Responsible Party: Sponsor-Investigator, Lu KZ, Southwest Hospital, Southwest Hospital, China
Organization: Southwest Hospital, China (Other)
Other Study IDs: LKZ-GAHBV-01
Record Dates: First submitted 2014-01-13; First posted 2014-01-16 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: HBV Infection
Keywords: Need general anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Days
Biospecimen Retention: Samples With DNA — serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- A: intravenous inhalational anesthesia
- B: intravenous anesthesia

SUMMARY:
The purpose of this study is to determine whether the general anesthesia immunosuppressive could effect hepatitis B Virus replication

DETAILED DESCRIPTION:
The change of immune state can influence HBV replication or elimination, it has been reported that a certain degree of immunosuppression occured after general anesthesia. In this study we detect the cytotoxic T lymphocyte(CTL) count and activity, interferon-γ(IFN-γ) and HBV-DNA content form the HBV patient who will accept general anesthesia. Our purpose is to evaluate the influence of general anesthesia immunosuppressive on HBV replication. If the results show that HBV-DNA quantity increases, so the patients might be given anti-HBV drugs or immune enhancer; otherwise it is indicated the general anesthesia immunosuppressive don't influence HBV replication.

ELIGIBILITY:
Inclusion Criteria:

1. American Society of Anesthesiologists（ASA） Ⅰ - Ⅱ;
2. ability to compliance the research plan;
3. volunteered and signed for the study ;
4. HBsAg positive, no serious system disease (heart: New York Heart Association（NYHA） class Ⅰ - Ⅱ, lung: vital capacity（VC）% or maximal voluntary ventilation（MVV）%>71, forced expiratory volume at one second（FEV1.0）%>61, arterial oxygen saturation（SaO2）%>94, arterial partial pressure of oxygen（PaO2）>75 mmHg, arterial carbondioxide partial pressure（PaCO2）<45mmHg, liver:child-pugh class A - B and kidney: chronic kidney disease（CKD）stage 1-3);
5. receive under general anesthesia (including gynecology, orthopedics,general surgery and urology department).

Exclusion Criteria:

1. ASA>Ⅱ;
2. tumor patients
3. can't collaborate;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with HBV infection receive surgery under general anesthesia
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2014-08 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
HBV-DNA | with in the first 5 days after surgery
  collect blood samples 4 times with in the first 5 days after surgery:
  the first time：before initiation of anesthesia; the second time：the first day after surgery; the third time：the third day after surgery; the forth time：the fifth day after surgery.
  And outcome measure will be assessed with in 3 months when all the samples collected, and will be presented with in 2 months when outcome measure assessed .

CONTACTS AND LOCATIONS:
Overall Officials: Lu KZ, PhD, Study Director — Department of Anesthesiology, Southwest Hospital Third Military Medical University
Locations (1):
- Department of Anesthesiology, Southwest Hospital Third Military Medical University, Chongqing, Chongqing Municipality, China

REFERENCES:
- [Derived] Quan J, Chen X, Tang X, Liu X, Li J, Yi B, Li P, Lu K, Gu J. Effects of General Anesthesia on Changes of Serum Hepatitis B Virus-DNA Levels in Infected Patients Underwent Non-Hepatobiliary Minimally Invasive Surgery: A Pilot Observational Study. Infect Drug Resist. 2022 Nov 11;15:6631-6640. doi: 10.2147/IDR.S379350. eCollection 2022. PMID 36386418